CLINICAL TRIAL: NCT06452329
Title: Retrospective Evaluation of Nivolumab in First-Line Unresectable Advanced or Metastatic Gastric Cancer (GC) and Gastroesophageal Junction Cancer (GEJC): A Non-interventional Observational Study in China
Brief Title: A Study to Evaluate Nivolumab in Patients With Unresectable Advanced/Metastatic Gastric Cancer and Gastroesophageal Junction Cancer
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-1429
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Participants who received first-line nivolumab therapy for advanced GC/GEJC
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — As prescribed by treating physician

SUMMARY:
The purpose of this study is to collect and evaluate real-world data to enhance understanding of the effectiveness, and treatment patterns of first-line nivolumab treatment in patients with unresectable advanced or metastatic gastric cancer/gastroesophageal junction cancer (GC/GEJC) in China

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥ 18 years at date of first administration of nivolumab
* Confirmed diagnosis of unresectable advanced or metastatic Gastric Cancer (GC) or Gastroesophageal Junction Cancer (GEJC) (histologically or cytologically)
* Participants newly received nivolumab as first-line (1L) treatment between 15 June 2018 and 30 June 2023
* Participants with at least one tumor assessment after index date except for death or discontinuation due to Adverse Events

Exclusion Criteria:

* Participants with primary malignancies other than unresectable advanced or metastatic GC/GEJC
* Participants who participate in an interventional clinical trial in or before 1L nivolumab treatment for advanced/metastatic GC/GEJC
* Participants with known HER2 status positive
* Participants who investigator deems inappropriate for inclusion, for example clinical data was incomplete

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with unresectable advanced or metastatic Gastric Cancer (GC) or Gastroesophageal Junction Cancer (GEJC) treated with nivolumab as first-line treatment.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Time to progression (TTP) | Up to 68 months

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 68 months
Duration of response (DOR) | Up to 68 months
Participant socio-demographics | Baseline
Participant baseline clinical characteristics | Baseline
Participant treatment patterns | Up to 68 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- China (2):
  - Local Institution - 0001, Wuhan, Hubei
  - Tianjin Happy Life Technology Co., Ltd, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts